CLINICAL TRIAL: NCT03916783
Title: Suubi4Cancer: An Innovative Combination Intervention to Improve Access to Pediatric Cancer Services and Treatment Adherence Among Children Living With HIV/AIDS in Uganda
Brief Title: Suubi4Cancer: Improving Access to Pediatric Cancer Services and Treatment Adherence Among Children Living With HIV/AIDS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We implemented Aims 1 and 2, but did not have a sufficient sample size to carry out the clinical trial portion
Sponsor: Washington University School of Medicine (Other)
Collaborators: Uganda Cancer Institute (Other); National Cancer Institute (NCI) (NIH); Reach the Youth Uganda (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R21CA236531 (NIH); 1R21CA236531-01 (NIH)
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: HIV/AIDS; Cancer
Keywords: Suubi; Youth; Poverty; Economic Empowerment Interventions; Epidemiology; Access to Treatment Services; Treatment Adherence; Uganda
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Due to insufficient sample size, the intervention (Aim 3) was not implemented. The enrolment number specified is for Aim 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination intervention (Experimental): Selected families will be assigned to the treatment condition (delivered over 9 months) to receive BSC plus a family EE intervention comprising of a matched family development account (FDA) for health-related expenses, including transport to UCI, food/nutrition, and health insurance. Combined with the Family EE will be four sessions of Financial Literacy and Management (FL&M) and two sessions of cancer education. The sessions will be conducted over a 4-week period. The two cancer-specific education sessions will use UCI materials to address: 1) definitions of cancer, potential causes, signs and symptoms, and importance of cancer testing; 2) debunking cultural explanations for the causes of cancer and misconceptions (beliefs, values, norms and prevailing attitudes)regarding cancer that largely impede service use.
  *Due to insufficient sample size, the open clinical trial is not being conducted.
  Interventions: Behavioral: Combination intervention

INTERVENTIONS:
Behavioral: Combination intervention — The FDA will be a matched savings account held in the child's name with the parent or caregiver as the co-signer, in a financial institution registered by the Central Bank (Bank of Uganda). The account opened will be matched with money from the program up to a match cap of 72,000 Uganda shillings (an equivalent of $20) a month per family for the 9-month intervention period.
  The FDAs will be complemented with four sessions of Financial Literacy and Management (FL&M) and two sessions of cancer education conducted over a 4-week period. The two cancer-specific education sessions will use UCI materials to address: 1) definitions of cancer, potential causes, signs and symptoms, and importance of cancer testing; 2) debunking cultural explanations for the causes of cancer and misconceptions (beliefs, values, norms and prevailing attitudes)regarding cancer that largely impede service use.
  Other Names: Family Development Account + Education Sessions

SUMMARY:
This study will tailor and explore the short-term preliminary outcomes of an existing evidence-based Economic Empowerment (EE) Intervention, Suubi (Hope in Luganda -local Ugandan language), on access to pediatric cancer diagnosis, care, and treatment adherence among youth living with HIV (YLWHIV) with suspected cancers. The study will specifically address the following aims/research questions: Aim 1. Identify confirmed and suspected cancer cases in a cohort of >3000 HIV+ youth (ages 10-24) seen at 39 clinics in 5 districts heavily affected by HIV/AIDS in southern Uganda. Aim 2. Identify those lost to follow-up from the cohort in Aim 1 and determine reasons for loss to follow-up through qualitative interviews. 2.1. Identify those who have not returned to the clinic in ≥ 60 days (~2 months) from their expected return visit date. 2.2. Determine reasons for loss to follow-up or death. Aim 3. Conduct an open clinical trial to establish the feasibility and acceptability of the Suubi4Cancer intervention.

*Due to insufficient sample size, Aim 3 is not implemented.

DETAILED DESCRIPTION:
While cancer studies among YLWHIV in sub-Saharan Africa (SSA) are rare, available literature demonstrates that HIV+ children have a greater risk for cancer (prior to antiretroviral therapy (ART)- >40-fold higher; post-ART- 4-14-fold higher) than their uninfected peers. Although ART is available to all Ugandan HIV+ children, only 47% were on ART in 2016. Additionally, some of the worst pediatric cancer survival rates worldwide are in SSA, with the majority dying from their disease. These dismal odds are influenced by several barriers to accessing cancer services and staying in treatment, including cultural misconceptions about cancer, and inadequate patient/family level resources. Based on our prior study findings among YLWHIV and informed by Asset theory, the investigators hypothesize that the main barriers to uptake of available cancer diagnostic testing, care and treatment adherence are financial and that through increased household and financial stability, the investigators can improve engagement with the health care system and seeking cancer care when confronted with a possible diagnosis.

Therefore this study is significant because the investigators will:

Aim 1. Identify confirmed and suspected cancer cases in a cohort of >3000 HIV+ youth (ages 10-24) seen at 39 clinics in 5 districts heavily affected by HIV/AIDS in southern Uganda

Aim 2. Identify those lost to follow-up from the cohort in Aim 1 and determine reasons for loss to follow-up through qualitative interviews.

2.1. Identify those who have not returned to the clinic in ≥ 60 days (~2 months) from their expected return visit date.

Approach: We will identify lost to follow-up individuals who in consultation with clinics government guidelines, and our records. We will exclude those with a reported vital status of the dead where it can be determined that they died of a condition other than possible cancer. We will also exclude those identified as having transferred to another clinic (also referred to as transfer outs), although, if well-documented, efforts will be made to track them and find out whether they are visiting the clinics/health care centers where they may have transferred to.

2.2. Determine reasons for loss to follow-up or death.

Approach: From those identified as lost to follow-up in 2.1, we will extract names, sex, birth date, and contact information including addresses, phone numbers, caregiver information, and clinic id. We will engage an expert client at each clinic to assist us with tracing of these individuals or their caregiving families for those documented as deceased where cancer/suspected cancer for child/youth was reported or no cause for death was reported. We will conduct in-depth interviews to determine reasons for not returning to HIV care, if not available from existing records and/or clinic personnel.

For those with phone numbers, we will contact them by telephone to tell them about the study and to determine if they are interested in participating. We will invite them to the clinic to present the study and allow them adequate time to consider whether or not they want to participate. If they participate, we will arrange to meet them to interview them for the study following consent.

For those without phone numbers, we will contact via expert clients available at each clinic, who will assist us with tracing of the individuals and inviting them for an introductory meeting to take place either at the clinic/healthcare center, in ICHAD's private research field offices in Masaka; or at the participants' homes (if they request it and there is sufficient privacy to ensure confidentiality). Flexibility in location when re-engaging and interviewing participants has been critical to our ICHAD studies success to date, including Suubi+Adherence whose infrastructure the current studies builds on.

Traced participants will be asked whether they are interested in participating in the study. We will provide them with a consent form (for caregivers) and assent forms for any child below 18 years of age.

Interviews determining reasons for lost to follow-up will focus on 1) experiences around HIV care at the clinic where they were a patient; 2) multi-level facilitators and barriers to access care; and 3) multi-level facilitators and barriers to staying in treatment.

2.3. For those determined to have died of cancer or with a suspected cancer identified from lost to follow-up interviews and from medical record abstraction for Aim 1, we will conduct the same interview as in 2.2 with additional questions with them or their identified primary caregiver to determine barriers and facilitators to cancer care.

- More specifically, the interviews will focus on1) experiences with their healthcare provider on communication around suspected cancer, and referral process; and 2) experiences with accessing services for further cancer testing, including barriers and facilitators to access

Aim 3. Conduct an open clinical trial to establish the feasibility and acceptability of the Suubi4Cancer intervention.

For cases identified with suspected cancers to date as a part of Aim 1 activities (n=7), those that are eligible will be invited to participate in an open clinical trial testing an economic empowerment intervention (Suubi4Cancer) to determine feasibility and acceptability.

We will conduct qualitative interviews to explore participants' experiences with the intervention, including feasibility and acceptability.

*Due to insufficient sample size, Aim 3 is not implemented.

ELIGIBILITY:
Inclusion Criteria:

Youth inclusion criteria are:

* HIV+ (confirmation by medical report)
* Must be living within a family (defined broadly, not necessarily with biological parents);
* Must be between 10-24 years old
* Attending one of the 39 clinics
* Did not access services or expressed unwillingness and/or inability to do so.

  * For Aim 1, inclusion criteria only includes 1) and 3).

Caregiver inclusion criteria:

* Have a YLWHIV (with suspected cancer) under their care who attends one of the 39 study-affiliated clinics.

Exclusion Criteria:

Potential participants will be excluded from the study if the research team determines that the participant:

* Cannot comprehend the study and participant rights
* Is unwilling to participate.

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Cancer Treatment Access | Every assessment time point (Baseline and at 9-month post-intervention initiation)
  Change in mean count of cases accessing cancer services.
Cancer Treatment Adherence | Every assessment time point (Baseline and at 9-month post-intervention initiation)
  Change in mean count of youth reporting adherence to prescribed cancer treatment.
Knowledge, Attitudes and Beliefs about Cancer and Cancer Treatment Services Composite measure | At 3-month post-intervention initiation (before and after the cancer education sessions)
  Change in knowledge, attitudes, and beliefs about cancer and cancer treatment services will be assessed by comparing pre- and post-study assessment questionnaire scores for participants in the intervention group. The assessment questionnaire is a composite measure developed for this study and adapted from several knowledge, attitudes and beliefs about cancer questionnaires including Attitudes and Beliefs about Cancer (ABC), Cancer Awareness Measure (CAM), Cancer Stigma Scale (CASS), and the Family CARE Project Baseline Questionnaire. The measure has a total of 13 questions ( including Yes- and No-types, questions on a scale of 1 (strongly agree) to 5 (strongly disagree) and descriptive questions such as health care provider preferences coded from 1 (medical doctor) to 4 (other)).

SECONDARY OUTCOMES:
Family and Social Support | Every assessment time point (Baseline and at 9-month post-intervention initiation)
  Change in family and social support. Family and social support will be assessed using the Social Support Behavior Scale (SS-B). The SS-B scale describes five central categories of supportive behaviors including emotional, socializing, practical, financial and advice/guidance which are assessed for both family and friends. The scale adapted for this study consists of 45 questions each with responses ranging from values of 1 (generally indicative of no support) to 5 (indicative of maximum support from both friends and family members). The theoretical range for this scale is 45-225, with higher scores indicating higher levels of social support from multiple sources.
Child Vulnerability in the Household index | Every assessment time point (Baseline and at 9-month post-intervention initiation)
  Change in child vulnerability in the household. Child vulnerability will be assessed using the Uganda Orphans and Vulnerable Children (OVC) Vulnerability Index (VI). This tool is intended for the selection of vulnerable households into OVC programs. The tool helps to determine a household's level of vulnerability (slight, moderate, and critical) based on individual and household level questions. The scale includes a total of 14 questions including descriptive questions for example; "Have you experienced any form of the following abuse in the last 30 days?" as well as nominal and ordinal-type questions, for example, questions whose responses are Yes- (labeled 0) and No-(labeled 4) as well as those ranked from 0 to 4, where a scale of four represents a greater vulnerability. The theoretical range for this scale is from 0 (lowest score - no vulnerability) to 56 ( highest score - high vulnerability). The higher the total score, the greater the child's vulnerability.
Savings Deposits | Every assessment time point (Baseline and at 9-month post-intervention initiation)
  Change in savings deposit.
Financial Literacy | Every assessment time point (Baseline and at 9-month post-intervention initiation)
  Increase in Financial Literacy knowledge. Participant knowledge of financial literacy will be assessed pre- and post- financial literacy sessions. The participants will be requested to respond to a series of 6 comprehensive questions to evaluate their attitudes towards saving. These questions include both descriptive and scale-type questions where participants will provide responses on a scale of 1 (Not important at all) to 5 (Extremely important) to statements about savings.
Intervention Feedback | At 9-month time point post-intervention initiation
  Semi-structured in-depth interviews will be utilized to obtain participants' feedback which will be utilized to inform future research with this population.
Intervention Satisfaction | At 9-month time point post-intervention initiation
  Client satisfaction surveys. The client satisfaction surveys will be utilized to assess participants' experiences with the intervention. The surveys will include a total of 8 questions, each with responses on a scale of 1 (No, definitely not) to 4 (Yes, definitely).

CONTACTS AND LOCATIONS:
Overall Officials: Fred M. Ssewamala, PhD, Principal Investigator — Washington University School of Medicine; Kimberly N Johnson, PhD, Principal Investigator — Washington University School of Medicine; Ozge Sensoy Bahar, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- International Center for Child Health and Development, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Once all of the data has been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community. The research team will make datasets available to any individual who makes a direct request to the PI and indicates the data will be used for the purposes of research (per CFR Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing, and evaluation, designed to develop or contribute to generalizable knowledge."). In sharing participant data, the team will follow Brown School at Washington University's Office of Sponsored Projects' data sharing agreements.
Time Frame: Will be determined on a case by case basis
Access Criteria: Will be determined on a case by case basis

REFERENCES:
- [Derived] Ssewamala FM, Sensoy Bahar O, Johnson KJ, Katumba RGN. Suubi4Cancer: A protocol for an innovative combination intervention to improve access to pediatric cancer services and treatment adherence among children living with HIV/AIDS in Uganda. Contemp Clin Trials Commun. 2019 Oct 1;16:100459. doi: 10.1016/j.conctc.2019.100459. eCollection 2019 Dec. PMID 31650077